CLINICAL TRIAL: NCT02655406
Title: COmpressioN Following Endovenous TreatmenT of Incompetent Varicose Veins (CONFETTI)
Brief Title: COmpressioN Following Endovenous TreatmenT of Incompetent Varicose Veins
Acronym: CONFETTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15/NE/0314
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Varicose Veins
Keywords: Foam sclerotherapy; Compression
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compression stockings (Active Comparator): Patients randomised to group A will be asked to wear compression stockings for 1 week
  Interventions: Other: Class 2 compression stockings
- No compression (No Intervention): Patients randomised to group B will be provided with bandages to wear for 24 hours only, with no further compression afterwards

INTERVENTIONS:
Other: Class 2 compression stockings
  Arms: Compression stockings

SUMMARY:
This study will be looking at the effect of compression therapy in patients having endovenous treatment for varicose veins using foam sclerotherapy. Patients will be randomised to either the compression group (group A) or the no compression group (group B).

The pain scores, compliance, quality of life scores, occlusion rate at 6 months as well as the cost effectiveness of each intervention will be assessed.

DETAILED DESCRIPTION:
This will be a randomised clinical trial looking at the impact of wearing or not wearing compression stocking following endovenous ablation using foam sclerotherapy.

Patients will be randomised to group A (compression) and group B (no compression).

Target Population Patients referred to the Imperial College NHS Trust for treatment of symptomatic varicose veins will be recruited if they are found to have varicose veins suitable for foam sclerotherapy on colour duplex scan.

Intervention

Patients will be randomised to have compression (group A) or no compression (group B). This will be done by using an online randomisation software (Sealed Envelope Ltd).

The compression therapy used will be Class II compression stockings. The treatment offered will be foam sclerotherapy of varicose veins using either Polidocanol or Sodium Tetradecyl Sulphate (STS) with the concentration used left to the discretion of the clinician.

Patients randomised to group A will be asked to wear compression stockings for 1 week.

Patients randomised to group B will be provided with bandages to wear for 24 hours only, with no further compression afterwards.

At baseline, patients will be asked to fill validated quality of life questionnaires (EQ-5D, AVVQ and CIVIQ) and will have their clinical scores assessed using a validated scoring system (CEAP and VCSS). On discharge after their varicose vein intervention, they will then be provided with a diary to record their post-procedural pain every day for 10 days using a validated visual analogue scale (VAS) as well as to record when they return to their normal activities and are back to work. They will also be asked to attend a follow-up in 2 weeks and at 6 months.

Patients' GP will also be sent a letter to inform them of their patient's participation in the study.

Follow-up

Patients will be followed up in the outpatient clinic at 2 weeks and 6 months.

Follow-up at 2 Weeks

At the 2 weeks' follow-up, the diary containing details of the pain scores and how soon patients were able to return to normal activities/work will be collected. In addition, patients will be asked about any phlebitis they have had in the two weeks after their procedure and how compliant they have been with the compression. They will be examined and the Venous Clinical Severity Score (VCSS) will be recorded. They will also be asked to fill in the EQ-5D, AVVQ and CIVIQ scores.

Follow-up at 6 Months

At the 6 months follow-up, patients will be examined and their VCSS will be recorded. They will also be asked to fill the EQ-5D, AVVQ and the CIVIQ scores. They will have a venous Duplex scan to determine occlusion of the treated vein.

Sample Size and Study Duration

We estimated the sample size needed to observe a difference of at least 10mm in the VAS score, with a standard deviation of 20mm. With power at 80% and 5% significance equivalence, we would need to recruit 128 patients (64 per group) to show a difference.

Previous studies looking at compression stockings have shown drop out rates close to 37% at 3 months10. Therefore, if we estimate a drop out rate of about 40% by 6 months, we would need to recruit at least 180 patients. If we recruit at least 2 patients per week, this will be approximately a total of 208 patients that could potentially be randomised over the course of two years.

With 6 months follow-up, therefore, the study will be running for 24 months with a target recruitment of 180 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Varicose veins suitable for foam sclerotherapy

Exclusion Criteria:

* Allergic to sclerosant
* Current DVT
* Arterial disease (ABPI<0.8)
* Patients unable to wear compression stockings
* Patients who are unwilling to participate
* Inability or unwillingness to complete questionnaires
* Inability to attend follow-up appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Patient's pain score post-procedure using a visual analogue scale (VAS) | 10 days
  Pain score

SECONDARY OUTCOMES:
Aberdeen Varicose Vein Questionnaire (AVVQ) score | 6 months
  Disease-specific quality of life score
Chronic venous insufficiency (CIVIQ) score | 6 months
  Disease-specific quality of life score
EuroQol's EQ-5D | 6 months
  Generic quality of life score
Venous clinical severity score (VCSS) | 6 months
  Clinical
Occlusion rate | 6 months
  Occlusion rates will be assessed based on a pre-agreed scale
Degree of phlebitis | 6 months
  Extent of phlebitis will be recorded using a scale

CONTACTS AND LOCATIONS:
Overall Officials: Roshan Bootun, Principal Investigator — Imperial College London
Locations (1):
- Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No